CLINICAL TRIAL: NCT07106021
Title: A Phase 1b/2a Study Assessing the Safety and Efficacy of Intraputamenal Dopaminergic Stem Cell Transplants in Patients With Idiopathic Parkinson's Disease
Brief Title: A Study to Assess Safety and Efficacy of Surgical Implant of RNDP-001 in Patients With Idiopathic Parkinson's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kenai Therapeutics (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RNDP-001-02
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Parkinson´s Disease; Parkinson's Disease
Keywords: RNDP-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (3):
- First patient group (Experimental): Low dose
  Interventions: Biological: RNDP-001; Device: Syringe Front-Loading Device
- Second patient group (Experimental): High dose
  Interventions: Biological: RNDP-001; Device: Syringe Front-Loading Device
- Third patient group (Experimental): Best dose
  Interventions: Biological: RNDP-001; Device: Syringe Front-Loading Device

INTERVENTIONS:
Biological: RNDP-001 — Stem cells
Device: Syringe Front-Loading Device — Delivers the stem cells

SUMMARY:
This clinical trial is designed to test the safety and tolerability of the study intervention, RNDP-001, which will be implanted into the brain of study participants during a surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease consistent with the Movement Disorders Society Clinical Criteria
* Age 45 to 75
* Medically stable to undergo a surgical procedure

Exclusion Criteria:

* Known Parkinson's disease gene mutation or variant
* Previous infusion therapy or surgery for Parkinson's disease
* History of allergic reaction or intolerance to an immunotherapeutic agent
* Contraindication to MRI
* Clinically significant medical conditions likely to interfere with the surgical procedure or study assessments

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline to 15 months post-transplant
  The incidence of adverse events (AEs), serious AEs, AEs of special interest, and patient withdrawals

SECONDARY OUTCOMES:
Changes from Baseline in Quality ON time measured by PD diary | Baseline to 15 months post-transplant
Changes in Dopaminergic Function and Activity in the Brain | Baseline to 15 months post-transplant
  Changes in L-DOPA-positron emission tomography (PET)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan will be determined later in the development.

REFERENCES:
- See also: Related Info — https://www.kenaitx.com/